CLINICAL TRIAL: NCT05126953
Title: 2-Hour Dispensing Evaluation of Samfilcon A Lenses With EPG01 Packaging Solution Compared to Commercially Available B+L Ultra Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-003
Record Dates: First submitted 2021-11-10; First posted 2021-11-19 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Contact Lens Wearer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Samfilcon A Lenses with EPG01 Packaging Solution (Experimental): Subjects implanted with Samfilcon A Lenses with EPG01 Packaging Solution
  Interventions: Device: samfilcon A Lenses with EPG01 Packaging Solution
- Commercially Available B+L Ultra Lenses (Active Comparator): Subjects implanted with Commercially Available B+L Ultra Lenses
  Interventions: Device: Commercially Available B+L Ultra Lenses

INTERVENTIONS:
Device: samfilcon A Lenses with EPG01 Packaging Solution — samfilcon A Lenses with EPG01 Packaging Solution
  Arms: Samfilcon A Lenses with EPG01 Packaging Solution
Device: Commercially Available B+L Ultra Lenses — Commercially Available B+L Ultra Lenses
  Arms: Commercially Available B+L Ultra Lenses

SUMMARY:
The objective of this 2 hour study is to evaluate the clinical performance of samfilcon A lenses with an alternate packaging solution (EPG01) compared to commercially available B+L Ultra lenses.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older on the date the Informed Consent Form (ICF) is signed and have capacity to read, understand and provide written voluntary informed consent.
2. Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
3. Have no active ocular disease or allergic conjunctivitis.
4. Not be using any topical ocular medications.
5. Be willing and able to follow instructions.
6. Have signed a statement of informed consent.

Exclusion Criteria:

1. Participating in a conflicting study in the opinion of the Investigator.
2. Considered by the Investigator to not be a suitable candidate for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Schafer, OD, Principal Investigator — Bausch & Lomb Incorporated
Locations (1):
- Bausch and Lomb Site 01, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a contralateral study. 30 subjects were enrolled and were dispensed lenses based on a randomization schedule.
Units Other Than Participants: Eyes
Groups:
- Samfilcon A Lenses With EPG01 Packaging Solution and Commercially Available B+L Ultra Lenses.: Each participant wore the test lens in one eye and the control lens in the fellow eye for 2 hours.
Period: Overall Study
Arm/Group | Samfilcon A Lenses With EPG01 Packaging Solution and Commercially Available B+L Ultra Lenses.
Started (30) | 30; 60 Eyes
Samfilcon A Lenses With EPG01 Packaging Solution | 30; 30 Eyes
B+L Ultra Lenses | 30; 30 Eyes
Completed | 30; 60 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Samfilcon A Lenses With EPG01 Packaging Solution and Commercially Available B+L Ultra Lenses.: Participants were implanted with both samfilcon A Lenses with EPG01 Packaging Solution and commercially available B+L Ultra lenses.
Arm/Group | Samfilcon A Lenses With EPG01 Packaging Solution and Commercially Available B+L Ultra Lenses.
Number analyzed (Participants) | 30
Number analyzed (Eyes) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.7 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Normalized logMAR Visual Acuity
Description: Normalized logMAR visual acuity is the change in visual acuity (how well you can see) from baseline (spectacle). Normalized visual acuity is calculated by subtracting the logMAR visual acuity with a contact lens from the baseline (refraction without a contact lens). Each letter on the logMAR visual acuity chart has a value of 0.02.
Time Frame: Assessed at 2-hour post-baseline
Measure: Mean (Standard Deviation); unit: LogMAR units
Units Other Than Participants: Lenses
Groups:
- Samfilcon A Lenses With EPG01 Packaging Solution: Participants were implanted with samfilcon A Lenses with EPG01 Packaging Solution
- Commercially Available B+L Ultra Lenses: Participants were implanted with commercially available B+L Ultra lenses.
Arm/Group | Samfilcon A Lenses With EPG01 Packaging Solution | Commercially Available B+L Ultra Lenses
Number analyzed (Participants) | 30 | 30
Number analyzed (Lenses) | 30 | 30
LogMAR units
  INS visit | 0.005 (0.0577) | 0.003 (0.0633)
  FUP visit | -0.001 (0.0663) | 0.008 (0.0632)

ADVERSE EVENTS:
Time Frame: Assessed at 2-hour post-baseline
Description: There were no adverse events with the samfilcon A lenses with EPG01 packaging solution.
  There were no adverse events with the commercially available. B+L Ultra lenses.
Groups:
- Samfilcon A Lenses With EPG01 Packaging Solution and Commercially Available B+L Ultra Lenses.: Participants wore samfilcon A lens with EPG01 in one eye and a commercially available B+L Ultra lens in the fellow eye
Arm/Group | Samfilcon A Lenses With EPG01 Packaging Solution and Commercially Available B+L Ultra Lenses.
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT05126953/Prot_SAP_000.pdf